CLINICAL TRIAL: NCT02723175
Title: The Effects of Cognitive Behavioral Therapy (CBT) and Transcranial Direct Current Stimulation (tDCS) on Fibromyalgia Patients
Brief Title: The Effects of CBT and tDCS on Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00039603; 1R21AR066428-01 (NIH)
Record Dates: First submitted 2015-12-14; First posted 2016-03-30 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-10

CONDITIONS: Fibromyalgia; Chronic Pain
Keywords: Fibromyalgia; Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham tDCS Stimulation (Experimental): 30 minutes of the sham transcranial Direct Current Stimulation
  Transcranial Direct Current Stimulation: Transcranial Direct Current Stimulation is a minimally invasive technique that uses a small amount of electricity (2mA) to temporarily stimulate specific brain areas in awake people.
  Interventions: Device: Transcranial Direct Current Stimulation
- Anodal tDCS Stimulation of DLPFC (Experimental): 30 minutes of the active transcranial Direct Current Stimulation (tDCS)
  Transcranial Direct Current Stimulation: Transcranial Direct Current Stimulation is a minimally invasive technique that uses a small amount of electricity (2mA) to temporarily stimulate specific brain areas in awake people.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation is a minimally invasive technique that uses a small amount of electricity (2mA) to temporarily stimulate specific brain areas in awake people.

SUMMARY:
Investigators are seeking to determine the effects of CBT, anodal tDCS over left DLPFC, and combined CBT+ tDCS on clinical pain and functioning among a sample of patients with fibromyalgia. This study will be the first randomized, double-blind, controlled study of tDCS technology as an adjunctive pain management strategy for fibromyalgia pain. Data from this trial will likely yield information regarding the feasibility and efficacy of tDCS+CBT as a chronic pain-management approach.

DETAILED DESCRIPTION:
Patients with fibromyalgia will complete questionnaires, six cognitive behavioral therapy sessions, quantitative sensory testing before and after the six therapy sessions, and undergo 30 minutes of tDCS during each of the six therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the American College of Rheumatology criteria for diagnosis of fibromyalgia for at least 1 year.
2. Between the ages of 21 and 85

Exclusion Criteria:

1. Other chronic pain conditions
2. on chronic opioid therapy
3. history of seizures
4. are or might be pregnant
5. metal/electronic implants or devices above the waist
6. moderate to severe depression (HDRS >19)
7. moderate to severe anxiety (BAI >16)
8. Latex allergy
9. Psychiatric illness other than mild depression or anxiety
10. on medications that lower seizure threshold

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Borckardt, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Started | 8 | 7
Completed | 4 | 4
Not Completed | 4 | 3
Not completed — Lost to 1 Month Follow Up | 3 | 2
Not completed — Lost to 3 Month Follow Up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.75 (10.25) | 48 (14.69) | 49.47 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Baseline Quantitative Sensory Testing (QST)
Description: Before treatment, Quantitative Sensory Testing (QST) will be completed for all participants. The QST involves a comprehensive laboratory pain assessment including heat stimuli using a Pathway Thermo-sensory Analyzer System which is specifically designed for assessing laboratory pain testing. The QST collects the temperature in celsius of when the participant first begins to feel the stimuli (Sensory), starts to feel pain (average pain threshold), and when the participant can no longer tolerate the stimuli (Tolerance). The temperature ranges from 37 degrees celsius to 50 degrees celsius. The minimum temperature on the scale is 37 degrees celsius and the maximum temperature on the scale is 50 degrees celsius. Average pain threshold: A lower temperature represents a lower pain threshold and a higher temperature represents a higher pain threshold. Tolerance: A lower temperature represents a lower pain tolerance and a higher temperature represents a higher pain tolerance.
Time Frame: Before Treatment
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 8 | 7
Degrees Celsius
  Sensory | 39.7063 (2.37354) | 39.8286 (1.85452)
  Average Pain Threshold | 43.9563 (3.19553) | 45.2036 (3.08134)
  Tolerance | 46.1531 (3.53357) | 47.2036 (2.24743)

2. Secondary Outcome: The Beck Depression Inventory (BDI) at Baseline
Description: The Beck Depression Inventory (BDI) will be used for screening purposes to characterize depression in each participant at baseline. The BDI is a 21 item participant rated inventory that evaluates depression symptoms, cognition, and physical symptoms of fatigue, weight loss, lack of interest in sex. The BDI scale also assesses suicidal ideation, those patients exhibiting suicidal ideations will be referenced to a therapist in order to further manage their depressive symptoms. The Total score range is 0 to 63; higher score indicates more depression. Individual items are scored on a 4 point scale (0 to 3), with 0=none/absent and 3=most severe.
Time Frame: Before Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 8 | 7
units on a scale | 21.38 (14.55) | 23.86 (11.82)

3. Secondary Outcome: The Beck Anxiety Inventory (BAI) at Baseline
Description: The Beck Anxiety Inventory (BAI) is a well-researched, brief self-report anxiety-screening instrument that assesses different aspects of anxiety experience (e.g., physiological, cognitive, behavioral). It was designed to measure participant's level of anxiety. The scale is unidimensional and the total score rages from 0 to 63. Low scores are associated with low levels of anxiety, while high scores are associated with high levels of anxiety.
Time Frame: Before Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 8 | 7
units on a scale | 12.75 (12.67) | 23.00 (11.33)

4. Secondary Outcome: Brief Pain Inventory-Average Pain at Baseline
Description: To assess each participant's average pain at baseline, the Brief Pain Inventory (BPI)-short form will be administered. The BPI rapidly assesses the severity of pain and its impact on functioning and has been widely used in both research and clinical settings. Participants rate their average pain in the past 24 hours using a 0-10 numerical rating scale, where 0=no pain and 10=extreme pain.
Time Frame: Before Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 8 | 7
units on a scale | 5.69 (2.39) | 7.06 (2.27)

5. Secondary Outcome: Percent Change in Average Daily Pain at Treatment Visit 3
Description: Participants were asked to rate their pain on average every day from the start of Treatment 1 until Treatment 3. Average pain ratings were on 0-10 scale. 0=No Pain at all and 10=Extreme Pain. Daily ratings were averaged at treatment 1 and treatment 3. The change in average daily pain ratings from treatment 1 to treatment 3 was calculated below. Time points at week 1 and week 3 were included to calculate percent change.
Time Frame: Treatment Session 3 (week 3)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 7 | 6
percent change | -13.29 (24.66) | -3.73 (12.64)

6. Secondary Outcome: Affective Subscale of McGill Pain Questionnaire at Baseline
Description: Participants completed the McGill Pain Questionnaire-short form (MPQ) at Baseline. The possible total range of scores (Sensory and Affective subscales together) is 0 to 45. The MPQ has two pain dimensions: 1.Sensory subscale awith 11 words, and 2.Affective subscale with 4 words from the original MPQ. The range of scores for the sensory dimension of pain is 0-33. The data below report the mean score for the affective subscale for both groups. The range of scores for the affective subscale being 0-12 with Higher scores indicating worse pain.
Time Frame: Before Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 8 | 7
units on a scale | 5.625 (3.24) | 6.714 (2.91)

7. Secondary Outcome: The Short-Form 12 Healthy Survey at Baseline
Description: To assess each participant's mental and physical functioning at Baseline, The Short-Form 12 Healthy Survey (SF-12) will be administered. The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey (Ware, Kosinski, and Keller, 1996). The questions were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. Total score range for the summary scores = 0-100, where higher score represents higher level of functioning.
Time Frame: Before Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 8 | 7
units on a scale | 30.13 (1.55) | 31.14 (2.73)

8. Secondary Outcome: The Fibromyalgia (FM) Impact Questionnaire at Baseline
Description: To assess the impact of fibromyalgia on each participant's function at baseline, The Fibromyalgia (FM) Impact Questionnaire will be administered. The FM assesses the following symptoms; physical Impairment, well-being, pain, fatigue, rested, stiffness, anxiety, and depression within the past 24 hours. Each symptom scale ranges from 0 to 10. For example, 0=no pain and 10=extreme pain, 0=not fatigued and 10=extremely fatigued. The final score is the total score which ranges from 0 to 80. Higher scores indicate greater impact of fibromyalgia on functioning.
Time Frame: Before Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 8 | 7
units on a scale | 3.46 (1.61) | 3.96 (0.79)

9. Secondary Outcome: The Beck Depression Inventory (BDI) at 1 Month Follow up
Description: The Beck Depression Inventory (BDI) will be used for screening purposes to characterize depression in each participant at the one month follow up visit. The BDI is a 21 item participant rated inventory that evaluates depression symptoms, cognition, and physical symptoms of fatigue, weight loss, lack of interest in sex. The BDI scale also assesses suicidal ideation, those patients exhibiting suicidal ideations will be referenced to a therapist in order to further manage their depressive symptoms. The Total score range is 0 to 63; higher score indicates more depression. Individual items are scored on a 4 point scale (0 to 3), with 0=none/absent and 3=most severe.
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 5 | 5
units on a scale | 15.40 (18.96) | 17.40 (13.69)

10. Secondary Outcome: The Beck Anxiety Inventory (BAI) at 3 Month Follow Up
Description: as for outcome 3
Time Frame: 3 Month Follow Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 4 | 4
units on a scale | 14.75 (23.09) | 16.75 (14.41)

11. Secondary Outcome: Brief Pain Inventory-Average Pain at 1 Month Follow Up
Description: At the one month follow up visit, The Brief Pain Inventory (BPI)-short form will be administered to assess each participant's pain on average in the past 30 days. The BPI rapidly assesses the severity of pain and its impact on functioning and has been widely used in both research and clinical settings. Participants rate their pain on average in the past 30 days using a 0-10 numerical rating scale, where 0=no pain and 10=extreme pain.
Time Frame: 1 Month Follow Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 5 | 5
units on a scale | 3.78 (3.21) | 3.53 (1.91)

12. Secondary Outcome: Percent Change in Average Daily Pain at Treatment Visit Six
Description: Participants were asked to rate their pain on average every day from the start of Treatment 3 until Treatment 6. Average pain ratings were on 0-10 scale. 0=No Pain at all and 10=Extreme Pain. Daily ratings were averaged at treatment 3 and treatment 6. The change in average daily pain ratings from treatment 3 to treatment 6 was calculated below. Time points at week 3, and week 6 were included to calculate percent change.
Time Frame: Treatment Session 6 (week 6)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 5 | 6
percent change | -24.17 (31.51) | -5.32 (16.28)

13. Secondary Outcome: Percent Change in Average Daily Pain at 1 Month Follow Up
Description: Participants were asked to rate their pain on average every day 30 days post treatment 6 (1 month follow up). Average pain ratings were on 0-10 scale. 0=No Pain at all and 10=Extreme Pain. The 30 Daily ratings (Post Treatment 6) were averaged and The change in average daily pain ratings from treatment 6 to the 1 month follow up (30 days post completion of treatment visit 6) was calculated below. Time points week 6, and the 1 month follow up were included to calculate percent change.
Time Frame: 1 Month Follow Up
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 5 | 5
percent change | -36.11 (29.33) | -23.71 (28.74)

14. Secondary Outcome: Percent Change in Average Daily Pain at 3 Month Follow Up
Description: Participants were asked to rate their pain on average every day for 60 days, post 1 month follow up visit. Average pain ratings were on 0-10 scale. 0=No Pain at all and 10=Extreme Pain. The 3 Month Follow Up included 60 Daily Pain ratings (Collected Post 1 Month Follow Up) that were averaged. The change in average daily pain ratings from the 1 month follow up (30 days post completion of treatment visit 6) to the 3 Month Follow Up (60 days post completion of the 1 month follow up visit) was calculated below. Time points 1 month follow up, and 3 month follow up were included to calculate percent change.
Time Frame: 3 Month Follow Up
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 4 | 4
percent change | -31.15 (42.72) | -48.93 (37.73)

15. Secondary Outcome: Affective Subscale of McGill Pain Questionnaire at 1 Month Follow Up
Description: Participants completed the McGill Pain Questionnaire-short form (MPQ) at Baseline. The possible total range of scores is 0 to 45. The MPQ has two pain dimensions: 1.Sensory subscale with 11 words, and 2.Affective subscale with 4 words from the original MPQ. The range of scores for the sensory dimension of pain is 0-33. The data below report the mean score for the affective subscale of the McGill Pain Questionnaire for both groups. The range of scores for the affective subscale being 0-12 with Higher scores indicating worse pain.
Time Frame: 1 Month Follow Up
Population: 3 Sham tDCS Participants dropped out leaving 5 total participants in Sham group.
  2 Anodal tDCS Participants dropped out leaving 5 total participants in Anodal group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 5 | 5
units on a scale | 4.2 (2.64) | 5.0 (3.29)

16. Secondary Outcome: The Short-Form 12 Healthy Survey at 1 Month Follow Up
Description: To assess each participant's mental and physical functioning at the 1 Month Follow Up visit, The Short-Form 12 Healthy Survey (SF-12) will be administered. The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey (Ware, Kosinski, and Keller, 1996). The questions were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. Total score range for the summary scores = 0-100, where higher score represents higher level of functioning.
Time Frame: 1 Month Follow Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 5 | 5
units on a scale | 29.60 (2.61) | 31.20 (1.92)

17. Secondary Outcome: The Fibromyalgia (FM) Impact Questionnaire at 1 Month Follow Up
Description: To assess the impact of fibromyalgia on each participant's function at the 1 Month Follow Up visit, The Fibromyalgia (FM) Impact Questionnaire will be administered. The FM assesses the following symptoms; physical Impairment, well-being, pain, fatigue, rested, stiffness, anxiety, and depression within the past 24 hours. Each symptom scale ranges from 0 to 10. For example, 0=no pain and 10=extreme pain, 0=not fatigued and 10=extremely fatigued. The final score is the total score which ranges from 0 to 80. Higher scores indicate greater impact of fibromyalgia on functioning.
Time Frame: 1 Month Follow Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 5 | 5
units on a scale | 3.31 (1.51) | 2.69 (1.23)

18. Primary Outcome: Post Baseline Quantitative Sensory Testing (QST)
Description: After treatment, Quantitative Sensory Testing (QST) will be completed for all participants. The QST involves a comprehensive laboratory pain assessment including heat stimuli using a Pathway Thermo-sensory Analyzer System which is specifically designed for assessing laboratory pain testing. The QST collects the temperature in celsius of when the participant first begins to feel the stimuli (Sensory), starts to feel pain (average pain threshold), and when the participant can no longer tolerate the stimuli (Tolerance). The temperature ranges from 37 degrees celsius to 50 degrees celsius. The minimum temperature on the scale is 37 degrees celsius and the maximum temperature on the scale is 50 degrees celsius. Average pain threshold: A lower temperature represents a lower pain threshold and a higher temperature represents a higher pain threshold. Tolerance: A lower temperature represents a lower pain tolerance and a higher temperature represents a higher pain tolerance.
Time Frame: One week Post Treatment
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
Number analyzed (Participants) | 5 | 6
Degrees Celsius
  Sensory | 39.2350 (3.53613) | 38.9083 (2.63726)
  Average Pain Threshold | 42.3050 (4.94057) | 44.1042 (4.10668)
  Tolerance | 44.1050 (5.50248) | 46.0417 (4.35634)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Sham tDCS Stimulation | Anodal tDCS Stimulation of DLPFC
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02723175/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-09-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT02723175/Prot_SAP_001.pdf